CLINICAL TRIAL: NCT06715943
Title: Multicenter, Single-arm, Open-label Phase III Study to Evaluate Efficacy and Safety of HRS-5965 Capsule in Patients With PNH Who Are Still Anemia After Anti-C5 Antibody Treatment
Brief Title: Efficacy and Safety of HRS-5965 in Patients With PNH Who Are Still Anemia After Anti-C5 Antibody Treatment
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chengdu Suncadia Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HRS-5965-302
Record Dates: First submitted 2024-11-28; First posted 2024-12-04 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Paroxysmal Nocturnal Hemoglobinuria
MeSH Terms: conditions — Hemoglobinuria, Paroxysmal

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HRS-5965 capsule (Experimental)
  Interventions: Drug: HRS-5965 capsule

INTERVENTIONS:
Drug: HRS-5965 capsule — HRS-5965 capsule treatment

SUMMARY:
This trial is a multi-center, single-arm, open-label phase III clinical trial. A total of approximately 35 patients with paroxysmal nocturnal hemoglobinuria who remained anemic despite stable use of C5 complement inhibitor (eculizumab/Kevacumab) for the first 6 months before randomization were included in the study. Approximately 40% of the subjects had received at least one red blood cell (RBC) transfusion within the first 6 months before receiving the experimental intervention. Subjects who met the criteria were all treated with HRS-5965 capsules. This trial includes an 8-week screening period, a 24-week treatment period, a 2-week dose reduction period, and a 4-week safety follow-up period.

ELIGIBILITY:
Inclusion Criteria:

1. Understand the specific process of the experiment, voluntarily participate in this experiment, and sign a written informed consent form.
2. Age ≥18 on the day of signing the informed consent, regardless of gender
3. It was confirmed to be PNH during screening, and the clone size of red blood cells or granulocytes was detected by flow cytopy >10%
4. Stable use of C5 complement inhibitor ikuzumab/covalimab for the first 6 months of random treatment
5. Have at least one blood transfusion record within the last 3 months, or sustain a hemoglobin level below 10g/dL during the eculizumab treatment within the last 3 months prior to screening.
6. The average hemoglobin level from two tests conducted by the central laboratory at the time of screening is less than 10 g/dL, with each individual Hb value being less than 10.5 g/dL.
7. Inoccution of Neisseris meningitis and Streptococcus pneumoniae vaccine at least 2 weeks before the first administration of HRS-5965; if HRS-5965 treatment must begin less than 2 weeks after vaccination, preventive antibiotic treatment must begin at least 2 weeks after vaccination.
8. Male and female subjects with fertility must agree to adopt efficient contraceptive measures with their partners within 30 days from the signing of the informed consent form to the last administration, and have no family planning and no sperm/egg donation.

Exclusion Criteria:

1. In addition to C5 complement inhibitors (ikuzuzumab/covalimamab), those who have participated in clinical trials of any other drug or medical device within 1 month before and are expected to have a residual effect of experimental treatment (judged by researchers), or those who were still in the follow-up period of a clinical trial or the 5 half-life of the experimental drug before screening Inside (whichever is longer)
2. Known or suspected hereditary or acquired complement deficiency
3. Currently active primary or secondary immunodeficiency
4. Those who have a history of splenectomy or plan to perform surgery during the trial
5. History of bone marrow/hematopoietic stem cells or solid organ transplantation
6. Diagnosed malignant tumors in the past 5 years
7. There is laboratory evidence for patients with bone marrow failure during screening
8. History of infection with pod bacteria (such as Neisseris meningitis, Streptococcus pneumoniae, etc.)
9. There is or is suspected of systemic active bacteria, virus or fungal infection 2 weeks before the first administration of HRS-5965 (according to the researcher's judgment)
10. Fever occurs within 1 week before the first administration of HRS-5965 (body temperature ≥38 ℃)
11. Human immunodeficiency virus (HIV) infection
12. Hepatitis B surface antigen (HBsAg) and hepatitis C antibody (HCVAb) are positive during screening, or abnormal liver function test during screening
13. Use any of the following drugs, unless there is a stable treatment plan before screening: a) erythropoietin (ESA), hypoxic-inducing factor proaminoyl hydroxylase inhibitor (HIF-PHI) or immunosuppressant for at least 8 weeks b) Systemic use of glucocorticoids (≤15 mg/day Prednisone or equivalent doses of glucocorticoids) at least 4 weeks c) Vitamin K antagonists (such as warfarin) have a stable international standardized ratio (INR) at least 4 weeks d) Low molecular weight heparin, oral anticoagulants such as aspirin, rvaroxaban, apifloxaban, etc. at least 4 weeks e) Iron supplements , vitamin B12, folic acid or androgen for at least 4 weeks
14. During screening, there are serious concurrent diseases, such as severe kidney disease (such as eGFR<30 mL/min/1.73 m2, dialysis), advanced heart disease (such as NYHA level IV), severe lung disease such as pulmonary hypertension (WHO level IV) or liver disease (such as active hepatitis), etc. , judged by the researcher that it is not suitable to participate in the researcher
15. Any medical condition determined by the researcher that it may affect the patient's participation in the trial, chronic anemia or unstable thrombosis events that may exist for other causes, and other conditions judged by the researcher to be unsuitable for participation in the trial
16. Those who are suspected of being allergic to experimental drugs or any ingredient in experimental drugs
17. Screening positive blood pregnancy test and breastfeeding women at the time of the visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2025-01-07 (Actual); Primary Completion 2026-01-06 (Actual); Study Completion 2026-01-06 (Actual)

PRIMARY OUTCOMES:
In the absence of red blood cell infusion (defined as no red blood cell infusion after week 2 to week 24), the proportion of subjects with at least 3 times of ≥12 g/dL of hemoglobin level measured 4 times between weeks 18 and 24. | From the 18th to the 24th week.

SECONDARY OUTCOMES:
The proportion of subjects who did not receive red blood cell infusion from week 2 to week 24 | From the 18th to the 24th week
The average change of hemoglobin compared with baseline during weeks 18 to 24 | From the 18th to the 24th week
The average percentage change of lactate dehydrogenase (LDH) level compared with the baseline during weeks 18 to 24 | From the 18th to the 24th week
The average change of reticular red blood cell count compared with the baseline during weeks 18 to 24 | From the 18th to the 24th week
Chronic Disease Treatment Function Assessment (FACIT) from weeks 18 to 24 - the average change of the score compared to the baseline | From the 18th to the 24th week
The incidence of breakthrough hemolysis from week 1 to week 24 | From the 18th to the 24th week
The incidence of MAVEs (including thrombosis) from week 1 to week 24 | From the 1st to the 24th week
The incidence and severity of adverse events from week 1 to week 24 | From the 1st to the 24th week
The concentration of HRS-5965 in plasma | From the 1st to the 24th week
The percentage of the change of complement bypass pathway (AP) activity at each point in time compared with the baseline | From the 1st to the 24th week

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Hematology Hospital of Chinese Academy of Medical Sciences, Tianjin, Tianjin Municipality
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: Undecided